CLINICAL TRIAL: NCT04022122
Title: Impact of Socio Economic Limitations on hEalth Outcomes in Patients With Complex and Advanced Chronic Cardiovascular Conditions in High-standard iNtegrated Care Environements (SELENE Study)
Brief Title: Impact of Socio Economic Limitations on Health Outcomes in Patients With Recent Admission for Heart Failure
Acronym: SELENE
Status: Completed | Type: Observational
Sponsor: Hospital Universitari de Bellvitge (Other)
Collaborators: Institut d'Investigació Biomèdica de Bellvitge (Other)
Responsible Party: Principal Investigator, Josep Comín, Head of the Cardiology Department and the Community Heart Failure Unit, Hospital Universitari de Bellvitge
Other Study IDs: IDIBELL-2019/PR157/19
Record Dates: First submitted 2019-07-14; First posted 2019-07-16 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Heart Failure
Keywords: Socioeconomic Level; Disease Management; Chronic Care Model; Transitional Care
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Heart Failure patients: The study does not imply any specific therapeutic intervention, and will not imply any change in the management of the participating patients, who will follow the usual clinical controls and will receive the medical and invasive treatments usually provided to patients with HF in our health area; as well as the different modalities of specific health education for this disease. At the time of hospital discharge, patients will be handled according to the usual protocols of the center established for outpatient follow-up of HF patients.
  Interventions: Procedure: Usual Care follow-up in a heart failure program.

INTERVENTIONS:
Procedure: Usual Care follow-up in a heart failure program. — Standard follow-up involves hospital and primary care for HF patients. In this context, physicians and nurses experienced in the care and management of HF direct care. HF care is based on 1) active detection of newly admitted HF patients, 2) planned educational interventions to improve self-care, 3) completion of a comprehensive psychosocial assessment of patients and caregivers, 4) discharge planning and home transition coordination involving the hospital HF team and Primary Care teams, 5) structured and planned evidence-based follow-up shortly after discharge from hospital.

SUMMARY:
To assess the impact of the socio-economic level on the effectiveness of a comprehensive multidisciplinary program of transitional care for crhonic heart failure patients (primary objective); to analyze this specifically in the various chronic management profiles of CHF patients and to study the associations between socio-economic level and other psychosocial aspects (secondary objective).

DETAILED DESCRIPTION:
The SELENE Study (Impact of SocioEconomic Limitations on health outcomes in patients with complex and advanced chronic cardiovascular conditions in high-standard iNtegrated care Environments) is an observational, cohort, prospective, multicenter study of consecutive patients treated in a comprehensive heart failure (HF) management program, and hospitalized by decompensated HF in our healthcare area; aimed at evaluating the impact of socioeconomic level on the effectiveness of a comprehensive multidisciplinary program of transitional care to patients with HF, both globally and in the various profiles of chronic management of HF.

In this study we aim to assess the impact of the socio-economic level on the effectiveness of a comprehensive multidisciplinary program of transitional care for chronic heart failure patients (primary objective); to analyze this specifically in the various chronic management profiles of HF patients and to study the associations between NSE and other psychosocial aspects (secondary objective).

All patients will have a detailed assessment by a social worker of a battery of psychosocial and functional variables, including educational level, functional status, cognitive status, family support, or the existence of a primary caregiver and an assessment of purchasing power through the value of monthly income. The events that will be analyzed, both for the primary objective of the study and the secondary objective related to the different follow-up profiles, will be re-admissions at 30 days (primary event), and mortality at 30, 90 and 180 days, as well as hospital admission at 90 days and 6 months (secondary events). Using the "median" income group as a reference, comparisons will be made between the rates of these events among the different groups.

The researchers hypothesize that the socioeconomic level has an impact on clinical events of HF patients so that the effectiveness of comprehensive care programs for HF is attenuated in patients with low socioeconomic level.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old.
* Patients discharged from a heart failure hospitalization within 30 days of enrollment into the study or in the process of discharge planning.
* Heart Failure diagnosis according to European Society of Cardiology (ESC) criteria.
* Written informed consent must be obtained before any assessment is performed.
* Patients receiving oral standard medication for chronic heart failure (CHF).
* All patients will be eligible regardless the level of left ventricular ejection fraction (LVEF).

Exclusion Criteria:

* Age<18 years old.
* Death before hospital discharge.
* The patient is unable or unwilling to give the informed consent to participate.
* Unstable patients with signs of fluid overload or low cardiac output.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: It will include, consecutively, all patients with a HF hospitalization within 30 days, discharged alive, and whose main diagnosis at discharge is HF.
Sampling Method: Non-Probability Sample
Enrollment: 121 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Occurrence of cardiovascular death or non-fatal heart failure events | Six months after inclusion of the patient.
  Occurrence of cardiovascular death or non-fatal heart failure events (time to first event) during a follow-up period of 6 months. Non-fatal heart failure event is defined as a new episode of worsening of symptoms and signs consistent with acute decompensated HF requiring intravenous decongestive therapy (e.g. diuretics) either on an outpatient basis (day-case HF hospital) or in the emergency department (<24 hours) or requiring unplanned hospital admission (>24 hours) or complicating the course of a non-cardiovascular admission.

SECONDARY OUTCOMES:
Readmission (all-cause, HF and cardiovascular) rate and total number. | Six months after inclusion of the patient.
  Comparison of the different socioeconomic levels at the end of follow-up.
Days in hospital (all-cause, HF and cardiovascular). | Six months after inclusion of the patient.
  Comparison of the different socioeconomic levels at the end of follow-up.
Rate of emergency visits. | Six months after inclusion of the patient.
  Comparison of the different socioeconomic levels at the end of follow-up.
Rate of non-fatal HF events. | Six months after inclusion of the patient.
  Comparison of the different socioeconomic levels at the end of follow-up.
Mortality for any cause and cardiovascular mortality. | Six months after inclusion of the patient.
  Comparison of the different socioeconomic levels at the end of follow-up.
Change of self-care using a validated scale (European Heart Failure Self-Care Behavior Scale) | Six months after inclusion of the patient.
  Comparison of the different socioeconomic levels at the end of follow-up.
Change of quality of life using a validated questionnaire (EUROQOL - 5D). | Six months after inclusion of the patient.
  Comparison of the different socioeconomic levels at the end of follow-up.
Patient satisfaction using a Likert-type scale. | Six months after inclusion of the patient.
  Comparison of the different socioeconomic levels at the end of follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Josep Comín Colet, MD,PhD, Principal Investigator — Head of the Cardiology Department and the Community Heart Failure Unit. MD, PhD
Locations (1):
- University Hospital Bellvitge, L'Hospitalet de Llobregat, Barcelona, Spain